CLINICAL TRIAL: NCT00516802
Title: A Phase I, Open Label, Study of the Safety and Tolerability of KU-0059436 and Dacarbazine in the Treatment of Patients With Advanced Solid Tumours
Brief Title: A Study to Assess the Safety and Pharmacokinetics of an Inhibitor of PARP in Combination With Dacarbazine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: KuDOS Pharmaceuticals Limited (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KU36-73; D0810C00003
Record Dates: First submitted 2007-08-13; First posted 2007-08-15 (Estimated); Last update posted 2009-05-15 (Estimated); Status verified 2009-05

CONDITIONS: Melanoma Neoplasms
Keywords: Poly(ADP ribose) polymerases; dacarbazine
MeSH Terms: interventions — olaparib; Dacarbazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): DTIC + KU-0059436
  Interventions: Drug: KU-0059436 (AZD2281)(PARP inhibitor); Drug: dacarbazine

INTERVENTIONS:
Drug: KU-0059436 (AZD2281)(PARP inhibitor) — oral
  Other Names: Olaparib
Drug: dacarbazine — intravenous injection over at least 20 minutes
  Other Names: DTIC

SUMMARY:
This is a Phase I, open-label, dose-escalating, study of the safety and tolerability of KU-0059436 in combination with DTIC in the treatment of patients with advanced melanoma who have not previously received systemic cytotoxic chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have:

  1. Unresectable stage 3 or stage 4 cutaneous melanoma or unknown primary melanoma with metastases.
  2. Histological or cytological confirmation of melanoma. Histological confirmation of melanoma from the primary site will suffice, unless the primary site is unknown.

Exclusion Criteria:

* Previous treatment with cytotoxic chemotherapy for advanced melanoma, apart from treatment for melanoma with isolated limb perfusion.
* Radiotherapy (except for palliative reasons), endocrine therapy, immunotherapy or use of other investigational agents within 4 weeks prior to trial entry (or a longer period depending on the defined characteristics of the agents used).
* Major surgery within 4 weeks of starting the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-01; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
To determine the safety, tolerability, dose-limiting toxicity (DLT), and (MTD) of KU-0059436 in combination with dacarbazine. | assessed every 3 weeks

SECONDARY OUTCOMES:
Objective tumour response | assessed every 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Prof James Carmichael, BSc MBChB MD FRCP, Study Director — KuDOS Pharmaceuticals Ltd; Prof Martin Gore, PhD MRCP FRCR, Principal Investigator — Royal Marsden Hospital Trust, London, UK
Locations (4):
- Research Site, Pittsburgh, Pennsylvania, United States
- United Kingdom (3):
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Oxford